CLINICAL TRIAL: NCT04105257
Title: Evaluation of Diagnostic Performance of Cerebral Perfusion Scans in Pseudo-Stroke: Exploratory Study of Diagnostic Performance
Brief Title: Evaluation of Diagnostic Performance of Cerebral Perfusion Scans in Pseudo-Stroke
Acronym: CTP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CE19.072
Record Dates: First submitted 2019-09-23; First posted 2019-09-26 (Actual); Last update posted 2022-12-12 (Actual); Status verified 2022-12

CONDITIONS: Stroke, Acute
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- All patients (Other): All patients seen at emergency with acute neurological deficit will be assessed if eligible to CTP/MRI
  Interventions: Diagnostic Test: All patients

INTERVENTIONS:
Diagnostic Test: All patients — Comparison of the results of the CTP with MRI

SUMMARY:
When a patient is received with the context of acute stroke, they undergo a fast neurological evaluation and obtain a basic appraisal composed of a non-contrast endovascular cerebral scan and an angiography scan of intracranial blood vessels and the neck. Once the structural lesion (hemorrhage, tumor, etc.) is absent, signs of early infracts and confirmed acute intracranial arterial occlusion, the possibility of a pseudo-stroke dwells in the differential diagnostic.

Certain characteristics of history and clinical evaluation create sufficient doubt to evoke the possibility of a pseudo-stroke. In fact, this population is mostly female and the cardiovascular risk factors are less prevalent in this group than for the group of stroke victims. It is on average the youngest and presents a less severe deficit. For the rest, medical antecedents often help to evoke a diagnosis of pseudo-stroke.

DETAILED DESCRIPTION:
With this study, the investigators wish to evaluate the diagnostic value of two additional radiological examinations:

1. Computed tomography perfusion (CTP) imaging to evaluate blood flow in the brain;
2. Imaging by magnetic resonance (MRI) of the brain to detect lesions from a cerebral vascular accident (stroke) not visible on standard imaging of the brain.

The proposed additional examinations (CTP and MRI) are tests that are currently used at the CHUM. Those are not experimental tests. These tests are commonly used when doctors wants a further investigation to clarify the cause of the neurological symptoms. These tests are usually done in a semi-urgent or non-urgent situations. In the present study they will be done urgently. The investigators wish to determine if obtaining these additional tests in emergency will change the decision of whether to administer the drug (thrombolysis). The investigators want to determine whether one imaging test is sufficient or if both exams are needed to help clinical decision-making. Please note that urgent access to perfusion CT and brain MRI is not considered routine care, since the value of these additional tests has yet to be demonstrated.

ELIGIBILITY:
Inclusion Criteria:

1. Admission at CHUM for acute neurological deficit <4,5h (since the onset of symptoms)
2. Potential candidate for an intravenous thrombolysis
3. Cerebral angioscan performed at CHUM at the time of admission
4. Age ≥ 18 years
5. Observed period from September 2019 à June 2020

Exclusion Criteria:

1. Contraindication to intravenous thrombolysis according to the doctor in charge of treatment;
2. Indication of a thrombectomy;
3. Incomplete exam or exam of insufficient technical quality for a reliable radiological interpretation;
4. Contraindication against MRI .

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2019-10-20 (Actual); Primary Completion 2022-10-04 (Actual); Study Completion 2022-10-04 (Actual)

PRIMARY OUTCOMES:
Sensibility | : Immediately after the procedure (CTP scan/MRI)
  proportion of patients that are correctly identified as having a pseudo-stroke
Specificity | Immediately after the procedure (CTP scan/MRI)
  proportion of patient that are correctly identified as not having a pseudo-stroke

CONTACTS AND LOCATIONS:
Overall Officials: Francois Guilbert, MD, Principal Investigator — Centre hospitalier de l'Université de Montréal (CHUM); Laura Gioia, MD, Principal Investigator — Centre hospitalier de l'Université de Montréal (CHUM)
Locations (1):
- Centre hospitalier de l'Université de Montréal (CHUM), Montreal, QC - Québec, Canada

IPD SHARING:
Plan to Share IPD: No